CLINICAL TRIAL: NCT06914817
Title: Brillouin Microscopy Used to Evaluate Corneal Mechanical Properties in Patients With Corneal Dystrophies and Post-Corneal Surgery: a Pilot Study
Brief Title: Brillouin Microscopy Used to Evaluate Corneal Mechanical Properties
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prim. Prof. Dr., Vienna Institute for Research in Ocular Surgery
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BMC
Record Dates: First submitted 2025-03-25; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Map Dot Fingerprint Dystrophy; Post-penetrating Keratoplasty; Post-Descemet Membrane Endothelial Keratoplasty; Healthy Corneas; Fuchs Endothelial Dystrophy; Ost-Descemet Stripping Automated Endothelial Keratoplasty
MeSH Terms: conditions — Corneal dystrophy, epithelial basement membrane; Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (8):
- Fuchs' Endothelial Dystrophy (FED) Group (Other)
  Interventions: Device: Brillouin optical scanning system (Intelon Optics) (BOSS)
- Map Dot Fingerprint Dystrophy (MDFD) Group (Other)
  Interventions: Device: Brillouin optical scanning system (Intelon Optics) (BOSS)
- Post-Penetrating Keratoplasty (PKP) Group (Other)
  Interventions: Device: Brillouin optical scanning system (Intelon Optics) (BOSS)
- Post-DSAEK Group (Other)
  Interventions: Device: Brillouin optical scanning system (Intelon Optics) (BOSS)
- Post-DMEK Group (Other)
  Interventions: Device: Brillouin optical scanning system (Intelon Optics) (BOSS)
- Pre- and Post-DSAEK Group (Other)
  Interventions: Device: Brillouin optical scanning system (Intelon Optics) (BOSS)
- Pre- and Post-DMEK Group (Other)
  Interventions: Device: Brillouin optical scanning system (Intelon Optics) (BOSS)
- Healthy Control Group (Other)
  Interventions: Device: Brillouin optical scanning system (Intelon Optics) (BOSS)

INTERVENTIONS:
Device: Brillouin optical scanning system (Intelon Optics) (BOSS) — Brillouin microscopy is a non-invasive optical imaging technique that measures the mechanical properties of tissues, such as stiffness and elasticity, by analyzing light scattering caused by natural acoustic waves within the tissue.

SUMMARY:
This study aims to explore the mechanical properties of the cornea using a non-invasive imaging technique called Brillouin microscopy. This innovative method measures corneal elasticity by detecting small shifts in light frequency, which occur due to interactions with acoustic waves in the tissue. These measurements can provide insights into how corneal stiffness is altered in various eye diseases or after surgery.

The study includes 100 participants, divided into different groups: patients with Fuchs' Endothelial Dystrophy (FED), Map Dot Fingerprint Dystrophy (MDFD), and those who have undergone corneal surgeries such as Penetrating Keratoplasty (PKP), Descemet's Stripping Automated Endothelial Keratoplasty (DSAEK), and Descemet Membrane Endothelial Keratoplasty (DMEK). Healthy individuals will also be studied as a control group.

Participants will first receive a standard eye exam, including a slit-lamp examination. Then, Brillouin microscopy will be used to measure the cornea's mechanical stiffness. Additional tests include optical coherence tomography (OCT), corneal topography and tomography, pachymetry (measuring corneal thickness), endothelial cell count, and intraocular pressure (IOP) measurement.

The purpose of this study is to better understand how diseases and surgeries affect corneal biomechanics. The researchers will also examine how well the Brillouin measurements match with findings from other clinical imaging tests. The results may help improve diagnosis and treatment options for corneal disorders.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to surgery
* Patients aged 18 years and older
* Patients who have undergone one of the following corneal surgeries or are diagnosed with one of the following dystrophies:

  * Penetrating Keratoplasty (PKP) and no longer have sutures following PKP o Descemet's Stripping Automated Endothelial Keratoplasty (DSAEK)
  * Descemet Membrane Endothelial Keratoplasty (DMEK)
  * Fuchs' Endothelial Dystrophy (FED)
  * Map Dot Fingerprint Dystrophy (MDFD)
* Healthy Controls: healthy eyes without any history of corneal diseases or surgeries

Exclusion Criteria:

Any of the following will exclude a subject from the study:

* Patients with inadequate corneal imaging or corneal scarring that would impact results
* Patients with other corneal dystrophies or corneal diseases
* Patients with active ocular infections or inflammatory conditions
* Patients unable to undergo Brillouin imaging adequately
* Patients that suffered an eye trauma according to their medical history
* Patients with fixational problems (e.g., head tremor) or with any medical condition that could interfere with the measurements
* Pregnancy (pregnancy test will be performed in women of reproductive age)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Brillouin shifts | 5 months
  This study aims to use Brillouin microscopy to compare corneal elasticity, measured in Brillouin shifts (GHz) among patients who have undergone corneal surgeries (PKP, DSAEK, DMEK), those with Map Dot Fingerprint Dystrophy (MDFD), and patients with Fuchs' Endothelial Dystrophy (FED).
  Outcome variables:
  * Correlation between Brillouin shifts in eyes post corneal surgery (PKP, DSAEK or DMEK) compared to healthy controls
  * Correlation between Brillouin shifts in eyes before corneal surgery compared to after corneal surgery (PKP, DSAEK or DMEK)
  * Correlation between Brillouin shifts in eyes with MDFD compared to healthy controls
  * Correlation between Brillouin shifts in eyes with FED compared to healthy controls

CONTACTS AND LOCATIONS:
Locations (1):
- VIROS - a Karl Landsteiner Institute, Vienna, Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vinciguerra R, Palladino S, Herber R, Romano MR, Vinciguerra P. The KERATO Biomechanics Study 1: A Comparative Evaluation Using Brillouin Microscopy and Dynamic Scheimpflug Imaging. J Refract Surg. 2024 Aug;40(8):e569-e578. doi: 10.3928/1081597X-20240701-02. Epub 2024 Aug 1. PMID 39120013